CLINICAL TRIAL: NCT02820766
Title: A Non-Randomized, Prospective Study of Short Term Outcomes Following Total Knee Replacement With JOURNEY™ II BCS Total Knee System Compared to Other Posterior Stabilized Total Knee Systems in a Physical Therapy Setting
Brief Title: Journey II BCS CMS Total Knee System Compared to Other PS Total Knee Systems in PT Setting
Status: Terminated | Type: Observational
Why Stopped: Logistics of study did not allow for consistent data collection
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Journey II BCS CMS Study
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis; Degenerative Arthritis; Traumatic Arthritis
Keywords: Posterior Stabilized Knee; Total Knee Arthroscopy; Journey II BCS
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Journey II BCS Knee: Physical Therapy Observational
- All Other Posterior Stabilized Knees: Physical Therapy Observational

SUMMARY:
The primary objective of the study is to determine how the short-term outcome of subjects implanted with the JOURNEY™ II BCS Total Knee System compares to subjects implanted with other PS total knee systems, and to determine if there is a difference in health care resources consumed that may result in economic savings to patients, the facility and/or the payer.

To address the study objectives, patient self-assessment questionnaires, and other objective measures of post-operative function and health care resource utilization will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Undergone unilateral primary total knee replacement with a JOURNEY™ II BCS Total Knee System or other Non-Smith & Nephew Posterior Stabilized Knee System
* Will be initiating outpatient PT ≤ 7 days post-operatively
* Has a primary diagnosis of osteoarthritis, degenerative arthritis, or traumatic arthritis
* Has pre-operative ROM ≥ 90°
* Is skeletally mature in the PI judgment
* Is 21 years of age of older
* Is willing and able to participate in required follow-up visits at the study site and to complete study procedures and questionnaires
* Has consented to participate in the study by signing the IRB/EC approved informed consent for the study
* Agrees to follow post- operative physical therapy program

Exclusion Criteria:

* Significant preoperative varus or valgus deformities (>15º)
* Has received a constrained or deep dish tibial insert
* Morbid obesity (BMI > 40)
* Has not obtained required pre-rehabilitation, pre-operative and intra-operative records by week 2 visit
* Other comorbidities that may impact outcomes such as osteoporosis, uncontrolled diabetes and active infection
* Fibromyalgia requiring treatment
* Current or impending incarceration or is a prisoner
* In the opinion of the PI has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse
* Is known to be at risk for lost to follow-up, or failure to return for scheduled visits
* Undergone or is planning to undergo total knee replacement of the contralateral knee within 6 months of this total knee replacement
* Requires a Legally Authorized Representative to consent to the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have a primary diagnosis of osteoarthritis, degenerative arthritis, or traumatic arthritis and who will receive either the Journey II BCS knee or any other posterior stabilized knee.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Difference in Knee Range of Motion (ROM) at the first outpatient Physical Therapy (PT) visit (≤7 days of surgery) between the 2 treatment groups | ≤7 days of surgery
  The absolute Range of Motion of index knee will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Beate Hanson, MD, Study Director — Smith & Nephew, Inc.
Locations (3):
- United States (3):
  - Anne Arundel Medical Cneter, Annapolis, Maryland
  - Slocum Research & Educational Foundation, Eugene, Oregon
  - University Orthopaedic Center, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Study terminated therefore no data sharing planned